CLINICAL TRIAL: NCT01986699
Title: Randomized Controlled Trial-Laparoscopic Assisted Colonoscopic Polypectomy
Brief Title: Laparascopic Assisted Colonoscopic Polypectomy
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Other Study IDs: 144467
Record Dates: First submitted 2013-10-29; First posted 2013-11-18 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Colon Polyps
Keywords: polypectomy; laparoscopic
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard Therapy: Patients are treated as per current standard of care
  Interventions: Procedure: Laparoscopic Assisted Polypectomy
- Laparoscopic Assisted Polypectomy: Patients treated with Laparoscopic Assisted Colonoscopic Polypectomy
  Interventions: Procedure: Laparoscopic Assisted Polypectomy

INTERVENTIONS:
Procedure: Laparoscopic Assisted Polypectomy

SUMMARY:
Study Objective: To compare the hospital costs between the standard surgical procedure and the Laparascopic Assisted Colonoscopic Polypectomy (LACP) technique for patients with advanced polyps in the colon.

DETAILED DESCRIPTION:
All patients being referred for possible LACP to the Division of Colorectal Surgery at Stony Brook University Medical Center will be randomized in a 1:1 fashion using a computer generated system to undergo either partial colectomy (performed by means of laparoscopy when possible), or LACP for the treatment of advanced polyp(s). Our research assistant will be present in the operating room to record the data.Patients will then undergo standard clinical management while hospitalized at Stony Brook according to the procedure performed.

ELIGIBILITY:
Inclusion Criteria:

* Polyp spanning 2 or more colonic folds
* Polyp > 20mm
* Polyp spanning greater than 50% of the colonic circumference
* Positive "lift sign" following submucosal injection of saline beneath the polyp
* Difficult location or position of the polyp, thus preventing assurance of complete endoscopic resection.

Exclusion Criteria:

* Polyps with histological evidence of adenocarcinoma
* Polyps in the rectum (<15cm from anal verge)
* Patients with known inflammatory bowel disease (IBD).
* Patients with known familiar adenomatous polyposis (FAP) syndrome
* Polyps without known histology (i.e. not previously biopsied)
* Polyps with large ulcerations, or those that demonstrate a "non-lift sign" during submucosal injection at the time of colonoscopy; as these are indicators of adenocarcinoma .
* Severe cardio-pulmonary disease, or irreversible coagulopathy, preventing abdominal surgery at an acceptable risk.
* POSSUM predicted mortality score greater than 2%
* Inability to obtain informed consent
* Patients under the age of 18
* Pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GI clinic
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
hospital cost | 1-3 days
  To compare the hospital costs between the standard surgical procedure and the LACP technique for patients with advanced polyps in the colon.

SECONDARY OUTCOMES:
complication rates | 1-3 days
  to compare complication rates between both techniques including intra-operative polypectomy related perforaton, polypectomy-related bleeding unable to be stopped endoscopically, post operative wound infection, ileus and anastomic leak.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto C Bergamaschi, MD, PhD, Principal Investigator — Stonybrook University
Locations (1):
- Stony Brook Medicine, Stony Brook, New York, United States